CLINICAL TRIAL: NCT05142527
Title: A Phase 2/3, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Safety, Tolerability, and Efficacy of ADM03820 to Prevent Symptomatic COVID-19 in Adult Subjects
Brief Title: Study to Evaluate the Safety and Efficacy of a Monoclonal Antibody Cocktail for the Prevention of COVID-19
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor withdrew study prior to initiation and no participants were enrolled.
Sponsor: Alachua Government Services, Inc. (Industry)
Collaborators: Enabling Biotechnologies (EB) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ADM03820-002
Record Dates: First submitted 2021-12-01; First posted 2021-12-02 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — ADM03820

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High Dose IM injection of active drug or Placebo (Phase 2) (Experimental): Subjects will receive a high dose IM injection of either active drug or placebo.
  Approximately 300 subjects will receive active drug and approximately 150 subjects will receive placebo in the Phase 2 segment.
  Interventions: Drug: ADM03820; Other: Placebo
- High Dose IM injection of active drug or Placebo (Phase 3) (Experimental): Subjects will receive a high dose IM injection of either active drug or placebo.
  Approximately 3000 subjects will receive active drug and approximately 1000 subjects will receive placebo in the Phase 3 segment
  Interventions: Drug: ADM03820; Other: Placebo

INTERVENTIONS:
Drug: ADM03820 — ADM03820 is a 1:1 mixture of two human IgG1 non-competitive binding anti-SARS-CoV-2 antibodies
Other: Placebo — Placebo

SUMMARY:
This is a Phase 2/3, randomized, double-blind, placebo-controlled, multi-center study to evaluate the safety, tolerability, and efficacy of ADM03820 to prevent symptomatic COVID-19 in adult subjects (≥ 18 years of age).

DETAILED DESCRIPTION:
Approximately 450 subjects will be enrolled in the Phase 2 segment of the study and will be randomized in a 2:1 ratio with a total of 300 subjects receiving ADM03820 and 150 subjects receiving placebo. In the Phase 3 segment, an additional 4,000 subjects will be enrolled and randomized in a 2:1 ratio, for a total sample size (including the Phase 2 subjects) of 4,450 total subjects.

The primary objective of the Phase 2 segment is to evaluate the safety and tolerability of ADM03820 in adult subjects. The secondary objectives are to assess safety, PK, immunogenicity, and microneutralization (MN) of ADM03820 and to gather information surrounding COVID-19 incidence rates and COVID-19 symptoms to support Phase 3 assumptions and assessment of efficacy.

The primary objectives of the Phase 3 segment are to evaluate the efficacy of ADM03820 for the prevention of symptomatic COVID-19 in adult subjects. The secondary objectives are to evaluate the efficacy of ADM03820 for prevention and amelioration of COVID-19 symptoms, to monitor the incidence and severity of COVID-19, and to evaluate the safety and tolerability of ADM03820.

ELIGIBILITY:
Phase 2 Inclusion Criteria:

1. Informed consent understood and signed prior to screening procedures
2. Healthy male or non-pregnant, non-lactating female 18 years of age or older, inclusive on the day of dosing
3. Subject willing to comply with and be available for all protocol procedures for the duration of the study
4. Subject determined by medical history, physical examination, and clinical judgement of the principal investigator (PI) to be eligible for inclusion in the study by meeting all the inclusion criteria and no exclusion criteria
5. Subject with BMI ≥18.5 and ≤ 35 kg/m2
6. Females of childbearing potential must have a negative urine pregnancy test on Day 1 prior to dosing Note: A woman is considered of childbearing potential unless post-menopausal (> or = 1 year without menses without other known or suspected cause and appropriately elevated FSH) or surgically sterilized via bilateral oophorectomy or hysterectomy.
7. Females of childbearing potential and males must agree to use medically effective contraception (methods with a failure rate of < 1% per year when used consistently and correctly) from screening until last dose. Acceptable methods include: hormonal contraception including implants, injections or oral; two barrier methods, e.g., condom and cervical cap (with spermicide) or diaphragm (with spermicide); intrauterine device or intrauterine system; abstinence when this is the subject's preferred and usual lifestyle.
8. Subject agrees to not donate bone marrow, blood, and blood products for at least 3 months after dosing
9. Clinical laboratory results within normal ranges or are no greater than Grade 1 and deemed not clinically significant by medical monitor and PI. (Any subjects with results that are Grade 2 or above according to toxicity table (modified from FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trial) will be excluded)
10. Subject willing to provide verifiable identification and has means to be contacted and to contact the Principal Investigator (PI) during the study.

Phase 2 Exclusion Criteria:

1. History of chronic medical condition that would either interfere with the accurate assessment of the objectives of the study or increase the risk profile of the subject
2. History of diabetes (type 1 or type 2), cardiovascular disease, pulmonary disease, chronic obstructive pulmonary disease (COPD) or asthma
3. History of severe allergic reactions of any type to medications, bee stings, food, or environmental factors or hypersensitivity or reaction to immunoglobins
4. Known allergic reactions or history of anaphylaxis or any other serious adverse reactions to any of the study product components present in the formulation or in its processing, as listed in the Investigator Brochure
5. Known to have HIV, HBsAg, or HCV per self-reported medical history
6. Febrile illness with temperature ≥38°C within 7 days of dosing. (Subjects with acute febrile illness within 7 days of dosing may be rescreened no earlier than 7 days following resolution of symptoms).
7. Rapid SARS CoV-2 antigen nasopharyngeal swab is positive on Day 1 prior to dosing or positive SARS-CoV-2 RT-PCR if result is received prior to dosing
8. Female subject who is pregnant or breastfeeding
9. Has previously received any coronavirus vaccine
10. Treatment with another investigational drug or licensed live vaccine within 30 days prior to or after planned enrollment. Subjects will be informed of local availability and be eligible to obtain an authorized COVID-19 vaccine at the time of enrollment and at any time during the study
11. Known history of COVID-19 infection
12. Receipt of any antibody (e.g. TIG, VZIG, IVIG, IM gamma globulin, monoclonal antibody) or blood or plasma transfusion within 6 months or within 5 half-lives of the specific antibody product given
13. History of solid organ or bone marrow transplantation
14. Active drug or alcohol use disorder or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
15. Use of H1 antihistamines or beta-blockers within 5 days of dosing (PRN use of H1 antihistamines may be acceptable after Medical Monitor approval)
16. History of malignancy within 5 years of screening (with the exception of squamous or basal cell carcinomas of the skin, or malignancy which is considered cured with minimal risk of recurrence)
17. Plans to enroll or is already enrolled in another interventional study
18. Has contraindication to IM injections or blood draws e.g., bleeding disorders, use of any anti-coagulants
19. Any specific condition that in the judgment of the PI precludes participation because it could affect subject safety
20. Is a study site employee or staff. Note: Site employees or staff include the PIs and sub-investigators or staff who are supervised by the PI or Sub-Investigators

Phase 3 Inclusion Criteria

1. Informed consent understood and signed prior to screening procedures
2. Healthy male or non-pregnant, non-lactating female 18 years of age or older, inclusive on the day of dosing
3. Subject has willingness to comply with and be available for all protocol procedures for the duration of the study
4. Subjects determined by medical history, physical examination, and clinical judgement of the PI to be eligible for inclusion in the study by meeting all the inclusion criteria and no exclusion criteria
5. Subject with BMI ≥18.5 and ≤ 40 kg/m2
6. Female subjects of childbearing potential must have a negative urine pregnancy test on Day 1 prior to dosing. Note: A woman is considered of childbearing potential unless post-menopausal (> or = 1 year without menses without other known or suspected cause and appropriately elevated FSH) or surgically sterilized via bilateral oophorectomy or hysterectomy
7. Females of childbearing potential must agree to use medically effective contraception (methods with a failure rate of < 1% per year when used consistently and correctly) from screening until last dose. Acceptable methods include: hormonal contraception including implants, injections or oral; two barrier methods, e.g., condom and cervical cap (with spermicide) or diaphragm (with spermicide); intrauterine device or intrauterine system; abstinence when this is the subject's preferred and usual lifestyle
8. Subject agrees to not donate bone marrow, blood, and blood products for at least 3 months after dosing
9. Subjects' willingness to provide verifiable identification, have means to be contacted and to contact the PI during the study

Phase 3 Exclusion Criteria:

1. History of chronic medical condition that would either interfere with the accurate assessment of the objectives of the study or increase the risk profile of the subject
2. History of severe allergic reactions of any type to medications, bee stings, food, or environmental factors or hypersensitivity or reaction to immunoglobins.
3. Known allergic reactions or history of anaphylaxis or any other serious adverse reactions to any of the study product components present in the formulation or in its processing, as listed in the Investigator Brochure
4. Febrile illness with temperature ≥38°C within 7 days of dosing. (Subjects with acute febrile illness within 7 days of dosing may be rescreened no earlier than 7 days following resolution of symptoms).
5. Rapid SARS CoV-2 antigen nasopharyngeal swab positive on Day 1 prior to dosing or positive SARS-CoV-2 RT-PCR if result is received prior to dosing
6. Female subject who is pregnant or breastfeeding
7. Treatment with another investigational drug or licensed live vaccine within 30 days prior to or after planned enrollment. Subjects will be informed of local availability and be eligible to obtain an authorized COVID-19 vaccine at the time of enrollment and at any time during the study
8. Known history of COVID-19 infection
9. Receipt of any antibody (e.g. TIG, VZIG, IVIG, IM gamma globulin, monoclonal antibody) or blood or plasma transfusion within 6 months or within 5 half-lives of the specific antibody product given
10. Active drug or alcohol use disorder or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
11. Plans to enroll or is already enrolled in another interventional study 12. Has contraindication to IM injections or blood draws e.g., bleeding disorders, use of any anti-coagulants
12. Has contraindication to IM injections or blood draws e.g., bleeding disorders, use of any anti-coagulants
13. Any specific condition that in the judgment of the PI precludes participation because it could affect subject safety
14. Is a study site employee or staff. Note: Site employees or staff include the PIs and sub-investigators or staff who are supervised by the PI or Sub-Investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of reactogenicity through Day 7 and adverse events (AEs) through end of study (Phase 2) | 540 days
  Number of participants with AEs and reactogenicity symptoms. FDA Toxicity Grading Scale for Local and General Systemic Reactogenicity will assess severity.
Incidence of SAEs and medically-attended AEs (Phase 2) | 540 days
  Number of participants with SAEs and medically-attended AEs through end of study
Occurrence of changes from baseline in physical examination, vital signs, and clinical safety laboratory values (Phase 2) | 365 days
  Number of participants with changes from baseline
Incidence of symptomatic, virologically confirmed COVID-19 (Phase 3) | Day 1 to Day 29
  Number of participants with symptomatic, virologically confirmed COVID-19

SECONDARY OUTCOMES:
Incidence of symptomatic, virologically confirmed COVID-19 (Phase 2 and Phase 3) | 183 days
  Number of participants with symptomatic, virologically confirmed COVID-19 through Day 183 (Phase 2) and through Day 57, Day 134, and Day 183 (Phase 3)
Hospitalization (Phase 2 and Phase 3) | 183 days
  Number of hospitalizations
All-cause mortality (Phase 2 and Phase 3) | 183 days
  Number of all-cause mortality
Incidence of AEs (Phase 2) | 540 days
  Number of participants with AEs through end of the study
Incidence of SAEs (Phase 2) | 540 days
  Number of participants with SAEs through end of the study
Incidence of COVID-19 related medically attended events (Phase 2) | 540 days
  Number of participants with events occurring after dosing through end of study
The assessment of Cmax for each of the monoclonal antibodies of ADM03820 as measured by mAb specific enzyme-linked immunosorbent assay (ELISA) (Phase 2) | 365 days
  Pre-dose and on Days 3, 8, 29, 57, 85, 134, 183, 232, 274 and 365
The assessment of Tmax for each of the monoclonal antibodies of ADM03820 as measured by mAb specific enzyme-linked immunosorbent assay (ELISA) (Phase 2) | 365 days
  Pre-dose and on Days 3, 8, 29, 57, 85, 134, 183, 232, 274 and 365
The assessment of AUC(0-t) for each of the monoclonal antibodies of ADM03820 as measured by mAb specific enzyme-linked immunosorbent assay (ELISA) (Phase 2) | 365 days
  Pre-dose and on Days 3, 8, 29, 57, 85, 134, 183, 232, 274 and 365
To assess SARS-CoV-2 antibody microneutralization levels (Phase 2) | 57 days
  Pre-dose and at Days 3, 29, and 57
To assess anti-drug antibody levels (Phase 2) | 365 days
  Pre-dose and on Days, 85, 134, 183, 232, 274, and 365
To assess daily COVID-19 symptoms (Phase 2) | 183 days
  COVID-19 daily symptoms reported by participants in diaries
SARS-CoV-2 RT-PCR assay in symptomatic subjects (Phase 2) | 540 days
Severity of each symptom (Phase 3) | 540 days
  Severity of symptoms are assessed from Day 1 through end of study
Incidence of mild, virologically confirmed COVID-19 (Phase 3) | 183 days
  Number of participants with mild, virologically confirmed COVID-19 through Days 29, 57, 134 and 183
Incidence of moderate, severe, or critical virologically confirmed COVID 19 (Phase 3) | 183 days
  Number of participants with moderate, severe, or critical virologically confirmed COVID 19 through Days 29, 57, 134, and 183
Incidence of and severity of virologically-confirmed COVID-19 (Phase 3) | 540 days
  Number of participants with virologically-confirmed COVID-19 and severity of symptoms from Days 29, 57, 134, and 183 through Day 540
Incidence of AEs, SAEs, and medically attended events (Phase 3) | 540 days
  Number of participants with AEs, SAEs, and medically attended events through end of study

OTHER OUTCOMES:
To assess Anti-SARS-CoV-2 Nucleoprotein (NP) antibody levels (Phase 2 and Phase 3) | 274 days
  Baseline and on Days 29, 57, 183 and 274
Serum collection for future analysis (Phase 2 and Phase 3) | 365 days
Collection of cDNA for SARS-CoV-2 sequence from subjects with positive RT-PCR assay (Phase 3) | 540 days

REFERENCES:
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300